CLINICAL TRIAL: NCT05595551
Title: Supporting Healthy and Sustainable Family Meals Among Parents With Lower Socioeconomic Status: Process and Effect Evaluation of the Project "Aan Tafel in 1,2,3 Euro"
Brief Title: Process and Effect Evaluation of the Project "Aan Tafel in 1,2,3 Euro"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2022-0343
Record Dates: First submitted 2022-10-17; First posted 2022-10-27 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Consumer Behavior; Food Selection
Keywords: Health promotion; Nutrition intervention; Socioeconomic status; Family meals; Parents
MeSH Terms: conditions — Consumer Behavior; Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention "Aan Tafel in 1, 2, 3 euro" (Experimental): The participants use the intervention program: the recipe booklets and the provided price guarantee for their meals.
  Interventions: Behavioral: The intervention "Aan Tafel in 1, 2, 3 euro"
- Control group (No Intervention): The participants are not registered to use the program and will be recruited in social organizations to match their sociodemographic profile as much as possible.

INTERVENTIONS:
Behavioral: The intervention "Aan Tafel in 1, 2, 3 euro" — The participants in this group are clients of Colruyt who are subscribed to the program "Aan Tafel in 1 2 3 euro". They will receive two-weekly recipe booklets with 6 balanced and child-friendly recipes in each booklet. They are guaranteed a fixed price for each recipe, that will be given at the checkout counter, based on their loyalty card.
  Arms: The intervention "Aan Tafel in 1, 2, 3 euro"

SUMMARY:
The goal of this research project is to learn what the impact of the specific project "Aan Tafel in 1 2 3 euro" is on the food and meal habits of families of lower SES.

Three types of studies will be conducted:

WP1) Process evaluation via qualitative research: focus groups and/or individual interviews with participants of Aan Tafel in 1 2 3 euro, and with delegates of the social organizations;

WP2) Effect evaluation via secondary data-analysis of purchase data retrieved from loyalty cards of participants, and of general customers (i.e., control group);

WP3) Process and effect evaluation with a control group in a baseline-post design: the intervention group are participants of the program, and the control group are clients in social organizations, but do not participate in the program.

On the one hand we want to find out if the intervention has an effect on specific determinants (i.e., food literacy, self-efficacy, attitudes, food security) of food behavior/meal prepping behavior and on meal structure of the family (i.e., amount of freshly made meals, amount of meals cooked and consumed together) (WP3), as well as on participants' food choices (WP2). On the other hand we want to find out how participans experience the program, what succes factors and barriers are, as well as how social organizations experience the program (as a partner of Colruyt, and contact person of the vulnerable families) (WP1).

DETAILED DESCRIPTION:
"Aan Tafel in 1 2 3 euro" is a project of retailer Colruyt in cooperation with social organizations in Belgium. The project/intervention was launched in 2016 and has been implemented throughout Belgium since. In 2021 about 8000 families have already been subscribed, and the numbers are still growing. Families with a lower SES (vulnerable families) are informed by a social organization (OCMW, CAW, kind & gezin, etc.) and can voluntarily register for the project. When a family is registered, they receive a recipe booklet every two weeks at home. The booklet consists of six easy, child-friendly recipes with accompanying shopping lists. Recipes are targeted at three people and include fish, meat and veggie dishes. Each recipe is guaranteed to cost no more than one, two or three euros per serving. The participants are registered via the Xtra-card (loyalty card of Colruyt), so that the discount can be offered anonymously and discretely. Since the intervention is an already existing one, we made an overview of the intervention components, behavior change techniques and practical applications, based on the Intervention Mapping Theory (Kok et al., 2015) and the Behavior Change Wheel (Abraham & Michie, 2008). Based on this overview, we determined goals and outcome measures for our research project.

In the qualitative study (WP1), participants of the intervention, as well as representatives of social organizations will be recruited to participate in an interview and/or focus group interview. Interviews will be conducted until data saturation is reached.

In the interventional study (WP3), participants of the project (intervention condition) will be compared to participants in a control condition who do not participate in the project. A total sample size of 200 participants is calculated, based on an a priori power analysis (two groups, two measurements, α=0.05; power=0.80, ES=0.25). Participants in both conditions will complete a survey in a pre-measurement and a post-measurement, three months after the start of the intervention.

The second effect study (WP2) has a longitudinal pre-post design, and is based on secondary purchase data from 2018 until 2022. The intervention group (i.e., participants of the intervention) will be compared to a control group (i.e., not subscribed in the intervention), by using general customer data. A multilevel growth model will be used to look at each individual's different purchase moments, with data before and during the intervention. The model represents three levels: 1) point of time/purchase, 2) customer, 3) store/location.

ELIGIBILITY:
Inclusion Criteria:

* Be registered for the project Aan Tafel in 1-2-3 euro
* Be a member of a family with at least one child under the age of 18 living at home.
* Being Dutch-speaking: thorough knowledge of Dutch in terms of reading/writing/speaking.
* Be over 18 years old and (regularly) responsible for the preparation of the family meals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Food literacy | Change from baseline food literacy at 3 months
  Food Literacy will be assessed via the 11 item questionnaire of Begley et al. (2018). And via the 6-item subscale 'Food preparation skills' of the Self-Perceived Food Literacy (SPFL) scale of Poelman et al. (2018).
Change in Self-efficacy for eating/cooking vegetables and fruits | Change from baseline self-efficacy at 3 months
  Self-efficacy will be measured with the 4-item subscale of the survey of Condrasky et al. (2011) 3. Food security, measured with the questionnaire of Gulliford et al. (2006)
Change in Cooking attitude | Change from baseline attitudes at 3 months
  Cooking attitudes will be measured with the 4-item subscale of the survey of Condrasky et al. (2011)
Change in Food security | Change from baseline food security at 3 months
  Food security will be assessed via the 18 Household Food Security Survey (HFSS) items of Gulliford et al. (2006)
Change in Family meal time frequency | Change from baseline meal time frequency at 3 months
  Family meal time frequency will be measured with an item out of the questionnaire of "Family meal time environment" of Fulkerson et al. (2006)
Change in Meal preparation | Change from baseline meal preparation at 3 months
  Meal preparation will be measured with an item out of the short questionnaire for assessing the impact of cooking skills interventions by Barton et al. (2011).
Change in food purchases (WP2) | Change from amount of food purchases before the subscription into the project at the time after subscription
  Food categories such as vegetables, ready-to-eat meals and snacks

SECONDARY OUTCOMES:
Change in Reported eating behavior | Change from baseline reported eating behavior at 3 months
  Specific food items related to mealtime are measured, based on the Health Behavior in School-aged Children (HBSC) survey.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Van Lippevelde, Study Director — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kok G, Gottlieb NH, Peters GJ, Mullen PD, Parcel GS, Ruiter RA, Fernandez ME, Markham C, Bartholomew LK. A taxonomy of behaviour change methods: an Intervention Mapping approach. Health Psychol Rev. 2016 Sep;10(3):297-312. doi: 10.1080/17437199.2015.1077155. Epub 2015 Oct 15. PMID 26262912
- [Background] Abraham C, Michie S. A taxonomy of behavior change techniques used in interventions. Health Psychol. 2008 May;27(3):379-87. doi: 10.1037/0278-6133.27.3.379. PMID 18624603
- [Background] Barton KL, Wrieden WL, Anderson AS. Validity and reliability of a short questionnaire for assessing the impact of cooking skills interventions. J Hum Nutr Diet. 2011 Dec;24(6):588-95. doi: 10.1111/j.1365-277X.2011.01180.x. Epub 2011 Jun 8. PMID 21649746
- [Background] Fulkerson JA, Neumark-Sztainer D, Story M. Adolescent and parent views of family meals. J Am Diet Assoc. 2006 Apr;106(4):526-32. doi: 10.1016/j.jada.2006.01.006. PMID 16567147
- [Background] Begley A, Paynter E, Dhaliwal SS. Evaluation Tool Development for Food Literacy Programs. Nutrients. 2018 Nov 2;10(11):1617. doi: 10.3390/nu10111617. PMID 30400130
- [Background] Poelman MP, Dijkstra SC, Sponselee H, Kamphuis CBM, Battjes-Fries MCE, Gillebaart M, Seidell JC. Towards the measurement of food literacy with respect to healthy eating: the development and validation of the self perceived food literacy scale among an adult sample in the Netherlands. Int J Behav Nutr Phys Act. 2018 Jun 18;15(1):54. doi: 10.1186/s12966-018-0687-z. PMID 29914503
- [Background] Condrasky MD, Williams JE, Catalano PM, Griffin SF. Development of psychosocial scales for evaluating the impact of a culinary nutrition education program on cooking and healthful eating. J Nutr Educ Behav. 2011 Nov-Dec;43(6):511-6. doi: 10.1016/j.jneb.2010.09.013. Epub 2011 Aug 15. PMID 21840764
- [Background] Gulliford MC, Nunes C, Rocke B. The 18 Household Food Security Survey items provide valid food security classifications for adults and children in the Caribbean. BMC Public Health. 2006 Feb 8;6:26. doi: 10.1186/1471-2458-6-26. PMID 16466571
- [Derived] Vos M, Proesmans VLJ, Van Kerckhove A, Deforche B, Michels N, Poelman MP, Van Lippevelde W. Evaluation of a national supermarket intervention supporting vulnerable families in healthy meal practices: a natural experiment. BMC Med. 2025 Jul 1;23(1):382. doi: 10.1186/s12916-025-04210-y. PMID 40597156
- [Derived] Vos M, Van Kerckhove A, Deforche B, Proesmans VLJ, Michels N, Poelman MP, Geuens M, Van Lippevelde W. Supporting vulnerable families' meal practices: process evaluation of a nationwide intervention implemented by a retailer and social organizations. BMC Public Health. 2024 Nov 6;24(1):3060. doi: 10.1186/s12889-024-20488-8. PMID 39506698